CLINICAL TRIAL: NCT05091021
Title: Skeletal Effects of Chronic Night Shift (ACORN Study)
Brief Title: Skeletal Effects of Chronic Night Shift
Acronym: ACORN
Status: Active, not recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-3014; R01HL151332 (NIH)
Record Dates: First submitted 2021-09-29; First posted 2021-10-25 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-05

CONDITIONS: Osteoporosis; Circadian Rhythm Sleep Disorder, Shift Work Type
MeSH Terms: conditions — Osteoporosis; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- University of Colorado Health New Nurses (Day Shift Workers): Day shift work group nurses have greater than 50% of their shifts as day shifts.
- University of Colorado Health New Nurses (Night Shift Workers): Night shift work group nurses have greater than 50% of their shifts as night shifts.

SUMMARY:
The specific aim of this observational study is to characterize changes in bone turnover makers (BTMs), bone mineral density (BMD), and bone microarchitecture in a cohort of nurses during their first year of night compared to day shift work. The hypothesis is that night shift nurses will have poorer bone health indices at one year compared to day shift nurses.

ELIGIBILITY:
Inclusion Criteria

* Healthy, nonpregnant adults 20-50 years old who recently (≤6 months) graduated from nursing school and were hired by University of Colorado Hospital for their first nursing position
* For women to be eligible, they must be premenopausal, not breastfeeding, not pregnant with no plans to become pregnant during the year of observation and willing/able to maintain their current method of contraception use as detailed below.
* Willing and able to travel to/from CU-AMC for study measurements at baseline and quarterly for one full year

Exclusion Criteria

* Non-nursing school related shift work 1 year prior to study. (note: many nursing students work as an Advanced Care Partner (ACP) or as a Student Nurse Extern (SNE) and these positions will not be considered exclusionary).
* Current smokers at baseline (or within the previous year of study).
* Individuals who are concurrently participating in another research protocol that would influence their safe participation in this study. For example, participants involved in a study that requires blood draws or ingestion of experimental medication as this would increase the risk of participation in our study and/or compromise study results.
* Any clinically significant unstable medical or surgical condition within the last year (treated or untreated), including history of a clinically significant abnormality of the neurological system (including cognitive disorders or significant head injury) or any history of seizure (including febrile seizure-sleep loss has been used clinically to induce seizures in patients with epilepsy). Given the wide range of illnesses that are encountered in medical practice, it would not be possible to provide a comprehensive list of each and every disease that could serve as grounds for exclusion for the subject. However, the following is a list of illness categories that would certainly be grounds for exclusion: Connective Tissue and Joint Disorders; Neurologic/cognitive Disorders; Musculoskeletal Disorders; Immune Disorders; Chronobiologic Disorders; Cardiovascular Disorders; Respiratory Disorders; Kidney Disorders; Infectious Diseases; Hematopoietic Disorders; Neoplastic Diseases; and Endocrine and Metabolic Diseases.
* Self-reported or newly diagnosed medical condition that is still being investigated or is not under good control, including those identified on screening labs such as:

  o Out-of-range values measured on a blood sample such as glucose, TSH, creatinine or hemoglobin, that represent clinically significant abnormalities that may jeopardize safe participation or accuracy of outcome measures, at PI discretion
* Any unstable psychiatric condition including but not limited to schizophrenic disorders and previously diagnosed personality disorders. Individuals with a history of anxiety or depression that has not required inpatient treatment and is well controlled without medication or on a stable medication dose will be permitted at the PI's discretion. Additionally, a personal history of limited prior counseling, psychotherapy (e.g., for adjustment reactions) will NOT be exclusionary.
* Evaluation of Psychiatric/Psychological Suitability:

  * Inability to demonstrate a full understanding of the requirements and demands of the study.
  * Individuals who are unaware of specific psychiatric diagnoses who have a history of having been treated with antidepressants, neuroleptic medications or major tranquilizers will be excluded from study.
* Individuals with any clinically significant sleep disorder; Diagnosis or symptoms of sleep disorders (history of significant parasomnia as an adult [night terrors, frequent sleep walking], insomnia, including but not limited to hypersomnias such as apnea, periodic limb movements, narcolepsy). Sleep disorders will be screened by self-report and physician interview including use of validated sleep questionnaires (PSQI, Epworth sleepiness scale, and Berlin sleep questionnaire for sleep apnea).
* Individuals on medications known to affect bone turnover (e.g., glucocorticoids, osteoporosis medications);
* Individuals with eGFR < 60 mL/min/1.73m2 as this is known to affect CTX measurements.
* Symptoms of active illness (e.g., fever) at time of enrollment; note - participant may be studied at a later date if they have not yet started their clinical duties by that time

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We will recruit volunteers from the pool of recently graduated new nurse hires at UCH. We will target our recruitment towards units that work the night shift (floor/ICU units) or day shifts (peri-operative and operating room units).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Difference in change of propeptide of type 1 procollagen (P1NP) over 1 year | From baseline up to 12 months
  Difference in change of P1NP over 1 year between the two groups (night vs. day shift nurses), as measured via bone biomarker assays (immunodiagnostic systems, chemiluminescence, immunoassay)

SECONDARY OUTCOMES:
Between-group differences in the change in osteocalcin | From baseline up to 12 months
  Between-group differences in the change in another bone formation marker (osteocalcin)
DXA-derived areal bone mineral density (aBMD) changes | From baseline up to 12 months
  Between-group differences in aBMD at the lumber spine, total hip and femoral neck measured by DXA
Change in bone microarchitecture | From baseline up to 12 months
  Change in trabecular volumetric BMD (vBMD) derived from high-resolution peripheral quantitative computed tomography (HR-pQCT)
Between-group differences in the change in CTX (C-telopeptide of type I collagen) | From baseline up to 12 months
  Between-group differences in the change in a bone resorption marker (CTX)

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Swanson, MD, MCR, Principal Investigator — CU Anschutz
Locations (1):
- CU Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No